CLINICAL TRIAL: NCT04322877
Title: Cardiac Resynchronisation Therapy In Patients With Heart Failure: Mechanistic Insights From Cardiac MRI And Electroanatomical Mapping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125230
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body surface mapping and temporary pacing (Experimental): Temporary pacing procedure with acute hemodynamic study and non-invasive body surface mapping.
  Interventions: Procedure: Temporary pacing Study; Radiation: Thoracic CT; Diagnostic Test: Acute hemodynamic study; Diagnostic Test: Non-invasive body surface mapping
- Catheter-based mapping and temporary pacing (Experimental): Temporary pacing procedure with acute hemodynamic study and invasive catheter-based mapping.
  Interventions: Procedure: Temporary pacing Study; Diagnostic Test: Acute hemodynamic study; Diagnostic Test: Invasive catheter-based mapping

INTERVENTIONS:
Procedure: Temporary pacing Study — Temporary delivery of CRT
  Other Names: Electrophysiology study
Radiation: Thoracic CT — As part of non-invasive mapping protocol
  Arms: Body surface mapping and temporary pacing
Diagnostic Test: Acute hemodynamic study — Measurement of invasive dP/dTmax
Diagnostic Test: Non-invasive body surface mapping — Cardioinsight body surface mapping
  Arms: Body surface mapping and temporary pacing
Diagnostic Test: Invasive catheter-based mapping — Invasive electroanatomical mapping
  Arms: Catheter-based mapping and temporary pacing

SUMMARY:
Cardiac Resynchronisation Therapy (CRT) is a specialist pacemaker procedure that aims to improve the efficiency of the heartbeat. This treatment is used routinely in patients with heart failure and a delay in electrical conduction across the heart seen on the surface ECG (heart tracing). The investigators aim to assess acute response to CRT and compare different methods of delivering CRT using hemodynamic data from invasive dP/dTmax and electroanatomical data from either invasive mapping or non-invasive body surface mapping.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Either 1) has CRT system in situ or 2) has a planned CRT system implant or 3) has a planned upgrade to CRT from a standard pacemaker
* NYHA grade II-IV heart failure
* LVEF<35%
* Intrinsic QRS duration >120ms
* On optimum medical therapy for heart failure
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participants who is pregnant, lactating or planning pregnancy during the course of the study.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Participant who is terminally ill or is inappropriate for placebo medication
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Rate uncontrolled atrial fibrillation precluding a cMR
* Significant peripheral vascular disease precluding an EP study
* A contraindication to anticoagulation
* A prosthetic aortic or tricuspid valve
* Significant Aortic valve disease
* Known LV thrombus
* Insufficient capacity to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in LV dP/dTmax >10 percent during temporary multisite pacing | Intra-procedure

SECONDARY OUTCOMES:
Electrical dyssynchrony measured from electro-anatomical mapping | Intra-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No